CLINICAL TRIAL: NCT00327288
Title: A Phase 1 Trial of Amplimexon® (Imexon, Inj.) Plus Taxotere® (Docetaxel) in Previously Treated Inoperable Stage III and Stage IV Non-Small Cell Lung Cancer (NSCLC), Locally Advanced or Metastatic Previously Treated Breast Cancer or Hormone Refractory Prostate Cancer
Brief Title: Safety Study of Imexon Plus Docetaxel in Lung, Breast or Prostate Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AmpliMed Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMP-010
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Non-small Cell Lung Cancer; Breast Cancer; Prostate Cancer
Keywords: Hormone refractory prostate cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Prostatic Neoplasms | interventions — 4-imino-1,3-diazabicyclo(3.1.0)hexan-2-one; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Docetaxel plus imexon
  Interventions: Drug: imexon; Drug: docetaxel

INTERVENTIONS:
Drug: imexon — IV variable dosages, days 1-5 every 21 days for duration of study
  Other Names: Amplimexon
Drug: docetaxel — IV once every 21 days for duration of study
  Other Names: Taxotere

SUMMARY:
Protocol AMP-010 is a Phase 1b study of imexon plus docetaxel for patients with previously treated breast cancer, previously treated lung cancer or hormone refractory prostate cancer. Docetaxel is approved by the Food and Drug Administration (FDA) as a second line therapy for these cancers. The imexon is administered on days 1-5 and the docetaxel on day 1 of every 3 week cycle. The objective of the protocol is to determine the highest dose of imexon which can be given with a full dose of docetaxel, and to provide information to enable the design of a future study focused on one or more specific cancer types.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with previously treated breast, lung, or prostate cancer where docetaxel is indicated.
* Prior treatment; at least one prior regimen required.
* Able to perform the activities of daily living.
* Off prior cancer therapy for at least 4 weeks.
* If female neither pregnant nor nursing.
* Willing to use contraceptives to prevent pregnancy.
* No other serious illnesses.
* No other active malignancy.
* No serious infections.
* No other current drug therapy for the cancer.
* Blood counts and blood chemistries in or near normal range.
* Prior radiation is permitted.

Exclusion Criteria:

* Active brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Determine the tolerability | duration of study
determine the maximally tolerated dose (MTD) | duration of study
determine the dose limiting toxicities (DLT) of increasing doses of imexon in combination with standard doses of docetaxel | duration of study
correlate changes in plasma glutathione (GSH) levels with imexon dose levels | cycle 1

SECONDARY OUTCOMES:
Record any objective tumor responses which may occur | duration of study

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site 008, Houston, Texas, United States

REFERENCES:
- [Result] Moulder S, Dhillon N, Ng C, Hong D, Wheler J, Naing A, Tse S, La Paglia A, Dorr R, Hersh E, Boytim M, Kurzrock R. A phase I trial of imexon, a pro-oxidant, in combination with docetaxel for the treatment of patients with advanced breast, non-small cell lung and prostate cancer. Invest New Drugs. 2010 Oct;28(5):634-40. doi: 10.1007/s10637-009-9273-1. Epub 2009 Jun 6. PMID 19499186